CLINICAL TRIAL: NCT01223300
Title: Osteoporosis Research Registry
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Thomas J. Schnitzer, professor, Northwestern University
Other Study IDs: STU00007523
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two (10 ml) blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Osteoporosis

SUMMARY:
The aim of this research registry is to collect information on individuals with osteoporosis, those with risk factors for osteoporosis, and comparative healthy controls. Bone mineral density measurements will be done on these individuals to determine bone health.

DETAILED DESCRIPTION:
The goal of this project is to develop a registry of research subjects with OP, with a risk of developing OP, and healthy controls. DXA scans will be performed on willing individuals at the spine, hips, and forearms and possibly the legs and heels in order to determine BMD. Subjects will also be asked to provide two (10 ml) blood samples, which may be used to analyze Vitamin D levels and/or other bone markers. By participating in the registry, subjects will be considered for current and future clinical research studies.

ELIGIBILITY:
Inclusion Criteria:

* Any subjects who give written informed consent

Exclusion Criteria:

* Any individual who is not willing or able to give written informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with osteoporosis or at risk for osteoporosis. Also, healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2008-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
BMD | 0 months

SECONDARY OUTCOMES:
Bone markers | 0 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Schnizter, M.D., PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States